CLINICAL TRIAL: NCT06599684
Title: Phase 2a Pilot, Open Label, Multicenter, Study of INV-102 Ophthalmic Solution in Subjects With Diabetic Macular Edema (DME) Associated With Non-proliferative Diabetic Retinopathy (NPDR)
Brief Title: Study of INV-102 Ophthalmic Solution in Adults With Diabetic Macular Edema Associated With Non-proliferative Diabetic Retinopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Invirsa, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INV-102-CS-004
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Non-center Involved Diabetic Macular Edema; Non-center Involved Diabetic Macular Edema Associated With Non-proliferative Diabetic Retinopathy; Diabetic Retinopathy; Center-involved Diabetic Macular Edema; Center-involved Diabetic Macular Edema Associated With Non-proliferative Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: INV-102 0.7% in NCIDME (Experimental): INV-102 0.7% Ophthalmic Solution given three times daily (TID) for 2 weeks followed by twice daily (BID) for 10 weeks
  Interventions: Drug: INV-102
- Part 2: INV-102 0.7% in CIDME (Experimental): INV-102 0.7% Ophthalmic Solution given three times daily (TID) for 2 weeks followed by twice daily (BID) for 6 weeks
  Interventions: Drug: INV-102

INTERVENTIONS:
Drug: INV-102 — 0.7% Ophthalmic Solution

SUMMARY:
Phase 2 study to assess the efficacy of topically administered eyedrops of INV-102 during a 12-week dosing period in subjects with non-center involved DME (NCIDME) associated with NPDR [Part 1] and during an 8-week dosing period in subjects with center-involved DME (CIDME) associated with NPDR [Part 2].

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female subjects ≥ 18 years of age and < 76 years of age
* Diagnosed with diabetes (Type 1 or 2) with hemoglobin A1c ≤ 12.0%
* Study eye must have NCIDME (Part 1) or CIDME (Part 2)
* Study eye must be moderate to severe NPDR

Key Exclusion Criteria:

* Prior laser treatment for DR in the study eye within 12 months from Screening Visit

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2024-09-07 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Early Treatment Diabetic Retinopathy (ETDRS) Diabetic Retinopathy Severity Scale (DRSS) score | Day 84 (Part 1) and Day 56 (Part 2)
  Graded by an independent central reading center using Wide-field Color Fundus Photography. The DRSS divides diabetic retinopathy into levels ranging from absence of retinopathy (score = 10) to advanced retinopathy (score = 85). The scale is used to describe overall retinopathy severity as well as the change in severity over time.
Change from baseline in central subfield thickness (Part 2 only) | Day 56
  Measured using spectral domain optical coherence tomography (SD-OCT) and determined by an independent central reading center.

SECONDARY OUTCOMES:
Change from baseline in macular volume | Day 84 (Part 1) and Day 56 (Part 2)
  Measured using spectral domain optical coherence tomography (SD-OCT)
Change from baseline in subfield thickness | Day 84 (Part 1) and Day 56 (Part 2)
  Mean retinal thickness in each of the regional subfields of the ETDRS grid, measured using SD-OCT
Change from baseline in the retinal thickness at the thickest point of the subfield thickness | Day 84 (Part 1) and Day 56 (Part 2)
  Measured using SD-OCT in each of the regional subfields of the ETDRS grid
Change in best corrected visual acuity (BCVA) (Part 2 only) | Day 56

CONTACTS AND LOCATIONS:
Overall Officials: Robert Shalwitz, Study Chair — Invirsa, Inc.
Locations (1):
- MedTrials, Inc., Dallas, Texas, United States